CLINICAL TRIAL: NCT04557215
Title: Evaluation of the Efficacy and Safety of Rifaximin in Combination With N-acetylcysteine (NAC) in Adult Patients With Irritable Bowel Syndrome With Diarrhea
Brief Title: Efficacy and Safety of Rifaximin With NAC in IBS-D
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Bausch Health Ireland Limited (Industry)
Responsible Party: Principal Investigator, Bianca Chang, GI Motility Clinic, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 550
Record Dates: First submitted 2020-09-11; First posted 2020-09-21 (Actual); Results first posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Irritable Bowel Syndrome With Diarrhea
Keywords: Irritable Bowel Syndrome with Diarrhea; IBS-D; Rifaximin; N-acetylcysteine; NAC
MeSH Terms: interventions — Rifaximin; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Standard dose for IBS-D (Active Comparator): Rifaximin 550 mg
  Interventions: Drug: Rifaximin
- Traveler's diarrhea dose + placebo (Placebo Comparator): Rifaximin 200 mg + placebo
  Interventions: Drug: Rifaximin; Drug: Placebo
- Traveler's diarrhea dose + NAC (Experimental): Rifaximin 200 mg plus N-acetylcysteine (NAC) 600 mg days
  Interventions: Drug: Rifaximin; Drug: N-acetylcysteine

INTERVENTIONS:
Drug: Rifaximin — Rifaximin is indicated for the treatment of irritable bowel syndrome with diarrhea (IBS-D) in adults.
  Other Names: xifaxan
Drug: N-acetylcysteine — N-acetylcysteine (NAC) is a clinically approved mucolytic agent.
  Other Names: NAC
  Arms: Traveler's diarrhea dose + NAC
Drug: Placebo — An inactive substance or treatment that looks the same as, and is given in the same way as, an active drug or intervention/treatment being studied.
  Arms: Traveler's diarrhea dose + placebo

SUMMARY:
Randomized, prospective proof of concept, double-blind, single site clinical trial to determine the efficacy of combined rifaximin and N-acetylcysteine (NAC) therapy vs. rifaximin alone in decreasing clinical symptoms in subjects with IBS-D.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is one of the most common functional gastrointestinal disorders, affecting 11% of the world's population, and accounting for 50% of all gastrointestinal office visits. IBS can be a chronic, long-term condition, with up to 57% of subjects who otherwise had normal bowel function continuing to have altered bowel function for at least 6 years after recovering from the initial acute illness. As a result, the health care costs of IBS have been estimated at over $30 billion per year. Further, this results in serious quality of life implications, which have been likened to diabetes or heart disease, in young adults who should otherwise be productive and healthy. IBS is characterized by abdominal pain, cramping and bloating, accompanied by altered bowel habits. The major forms of IBS are diarrhea-predominant (IBS-D), constipation-predominant (IBS-C) and mixed IBS (IBS-M).

There is significant bacterial involvement in IBS, particularly IBS-D. IBS-D can be precipitated by acute gastroenteritis, which is caused by infection with bacterial pathogens such as Escherichia coli, Salmonella, Shigella and Campylobacter jejuni. In addition, there is now overwhelming evidence that small intestinal bacterial overgrowth (SIBO) contributes to the symptoms of IBS-D. Therefore, antibiotic treatment has become a mainstay in the treatment of IBS. Of these, rifaximin is the only antibiotic currently approved by the FDA for the treatment of IBS-D. Rifaximin is an oral, broad-spectrum antimicrobial agent that is minimally absorbed (99.6% retained in the gut), targets the gastrointestinal tract, and associated with a low risk of clinically relevant bacterial antibiotic resistance. It is generally recognized as having no side effects in blinded comparisons that differ from placebo. In two identically designed, phase 3, double-blind, placebo-controlled trials of patients with IBS-D, 40.7% of patients treated with rifaximin 550 mg 3 times daily for 2 weeks experienced adequate relief of global IBS symptoms, compared with 31.7% of patients treated with placebo (P<0.001). In addition, a greater percentage of rifaximin-treated than placebo-treated patients reported durable improvement in IBS-D symptoms for at least 10 weeks post-treatment.

It is well known that treatment of IBS-D with rifaximin is effective and now FDA-approved. However, only 44% of subjects improved with rifaximin treatment. Although what is unique about rifaximin is its 'one-and-done' treatment effect, this is only seen in 36% of subjects who respond to this drug. As such, there is room for improvement with rifaximin. In recent studies, we have shown that the most predominant bacteria in the bacterial overgrowth associated with IBS are E. coli and Klebsiella. Rifaximin is highly effective in treating these two organisms. However, we have since learned that the majority of these excessive organisms in IBS are found in the small intestinal mucus layer. Since rifaximin is not soluble in mucus, it cannot penetrate and affect bacteria within the mucus layer. Our hypothesis that the addition of a mucolytic like N-acetylcysteine (NAC) will allow the penetration of rifaximin into the mucus by first solubilizing rifaximin and secondly liquifying the mucus. This may allow for two important effects. One is a reduction in the necessary dose of rifaximin necessary to treat IBS, and the other is improved efficacy. Both of these will be tested in this trial.

In this study, we propose to test whether combining rifaximin with a clinically approved mucolytic agent, NAC, can result in improvement in stool form and reduction in stool frequency, as well as improved relief of clinical symptoms, in subjects with IBS-D.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18-75 years old inclusive
* Onset of clinical symptoms for IBS-D occurring at least 6 months and, in order to progress to treatment phase, meet the following:

  1. Has abdominal pain, on average, ≥1 day per week in previous 3 months, associated with ≥2 of the following: (1) Related to defecation, (2) Associated with a change in stool frequency, or (3) Associated with a change in form (appearance) of stool.
  2. Fits Rome IV criteria for IBS with diarrhea (IBS-D), which is defined by >25% of abnormal bowel movements with Bristol stool form types 6 or 7 (loose, watery stool) and <25% of abnormal bowel movements with Bristol stool form types 1 or 2 (hard, lumpy stool).
* Colonoscopy must have been completed within the past 10 years
* Subjects are capable of understanding the requirements of the study, are willing to comply with all the study procedures, and are willing to attend all study visits
* All subjects (male and female) shall agree to use an acceptable method of contraception throughout their participation in the study. Acceptable methods of contraception include:

  1. Double barrier methods (condom with spermicidal jelly or a diaphragm with spermicide),
  2. Hormonal methods (e. g. oral contraceptives, patches or medroxyprogesterone acetate),
  3. An intrauterine device (IUD) with a documented failure rate of less than 1% per year.
  4. Abstinence or partner(s) with a vasectomy may be considered an acceptable method of contraception at the discretion of the investigator.
  5. Female subjects who have been surgically sterilized (e.g. hysterectomy or bilateral tubal ligation) or who are postmenopausal (total cessation of menses for >1 year) will not be considered "females of childbearing potential".

Exclusion Criteria:

* Use of any oral antibiotics in the last two months
* Subjects with history of intestinal surgery (except appendectomy or cholecystectomy)
* Subjects with known pelvic floor dysfunction
* Pregnancy
* Nursing mothers
* Poorly controlled/uncontrolled significant medical condition that would interfere with study procedures
* History of bowel obstruction
* History of inflammatory bowel disease or celiac disease
* History of HIV
* Cirrhosis
* IBS-C/chronic idiopathic constipation
* Poorly controlled diabetes or thyroid disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pimentel, MD, Study Director — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Johansson ME, Sjovall H, Hansson GC. The gastrointestinal mucus system in health and disease. Nat Rev Gastroenterol Hepatol. 2013 Jun;10(6):352-61. doi: 10.1038/nrgastro.2013.35. Epub 2013 Mar 12. PMID 23478383
- [Background] Ermund A, Schutte A, Johansson ME, Gustafsson JK, Hansson GC. Studies of mucus in mouse stomach, small intestine, and colon. I. Gastrointestinal mucus layers have different properties depending on location as well as over the Peyer's patches. Am J Physiol Gastrointest Liver Physiol. 2013 Sep 1;305(5):G341-7. doi: 10.1152/ajpgi.00046.2013. Epub 2013 Jul 5. PMID 23832518
- [Background] Oriano M, Terranova L, Teri A, Sottotetti S, Ruggiero L, Tafuro C, Marchisio P, Gramegna A, Amati F, Nava F, Franceschi E, Cariani L, Blasi F, Aliberti S. Comparison of different conditions for DNA extraction in sputum - a pilot study. Multidiscip Respir Med. 2019 Jan 31;14:6. doi: 10.1186/s40248-018-0166-z. eCollection 2019. PMID 30733864
- [Background] Leite GGS, Morales W, Weitsman S, Celly S, Parodi G, Mathur R, Sedighi R, Barlow GM, Rezaie A, Pimentel M. Optimizing microbiome sequencing for small intestinal aspirates: validation of novel techniques through the REIMAGINE study. BMC Microbiol. 2019 Nov 1;19(1):239. doi: 10.1186/s12866-019-1617-1. PMID 31675917
- [Background] Sadowska AM, Verbraecken J, Darquennes K, De Backer WA. Role of N-acetylcysteine in the management of COPD. Int J Chron Obstruct Pulmon Dis. 2006;1(4):425-34. doi: 10.2147/copd.2006.1.4.425. PMID 18044098
- [Background] Mokhtari V, Afsharian P, Shahhoseini M, Kalantar SM, Moini A. A Review on Various Uses of N-Acetyl Cysteine. Cell J. 2017 Apr-Jun;19(1):11-17. doi: 10.22074/cellj.2016.4872. Epub 2016 Dec 21. PMID 28367412
- [Background] Lembo A, Pimentel M, Rao SS, Schoenfeld P, Cash B, Weinstock LB, Paterson C, Bortey E, Forbes WP. Repeat Treatment With Rifaximin Is Safe and Effective in Patients With Diarrhea-Predominant Irritable Bowel Syndrome. Gastroenterology. 2016 Dec;151(6):1113-1121. doi: 10.1053/j.gastro.2016.08.003. Epub 2016 Aug 13. PMID 27528177
- [Background] Lovell RM, Ford AC. Global prevalence of and risk factors for irritable bowel syndrome: a meta-analysis. Clin Gastroenterol Hepatol. 2012 Jul;10(7):712-721.e4. doi: 10.1016/j.cgh.2012.02.029. Epub 2012 Mar 15. PMID 22426087
- [Background] Thompson WG. The functional gasterointestinal bowel disorders. In: Drossman DA, editor. The functional gaterointestinal disorders. Boston: Little, Brown; 1994. p. pp-117-134.
- [Background] Neal KR, Barker L, Spiller RC. Prognosis in post-infective irritable bowel syndrome: a six year follow up study. Gut. 2002 Sep;51(3):410-3. doi: 10.1136/gut.51.3.410. PMID 12171965
- [Background] The burden of gasterointestinal diseases. In: American Gastroenterological Association; 2001; Bethesda, MD; 2001.
- [Background] Lackner JM, Gudleski GD, Zack MM, Katz LA, Powell C, Krasner S, Holmes E, Dorscheimer K. Measuring health-related quality of life in patients with irritable bowel syndrome: can less be more? Psychosom Med. 2006 Mar-Apr;68(2):312-20. doi: 10.1097/01.psy.0000204897.25745.7c. PMID 16554399
- [Background] Okhuysen PC, Jiang ZD, Carlin L, Forbes C, DuPont HL. Post-diarrhea chronic intestinal symptoms and irritable bowel syndrome in North American travelers to Mexico. Am J Gastroenterol. 2004 Sep;99(9):1774-8. doi: 10.1111/j.1572-0241.2004.30435.x. PMID 15330917
- [Background] Mearin F, Perez-Oliveras M, Perello A, Vinyet J, Ibanez A, Coderch J, Perona M. Dyspepsia and irritable bowel syndrome after a Salmonella gastroenteritis outbreak: one-year follow-up cohort study. Gastroenterology. 2005 Jul;129(1):98-104. doi: 10.1053/j.gastro.2005.04.012. PMID 16012939
- [Background] Ji S, Park H, Lee D, Song YK, Choi JP, Lee SI. Post-infectious irritable bowel syndrome in patients with Shigella infection. J Gastroenterol Hepatol. 2005 Mar;20(3):381-6. doi: 10.1111/j.1440-1746.2005.03574.x. PMID 15740480
- [Background] Spiller RC, Jenkins D, Thornley JP, Hebden JM, Wright T, Skinner M, Neal KR. Increased rectal mucosal enteroendocrine cells, T lymphocytes, and increased gut permeability following acute Campylobacter enteritis and in post-dysenteric irritable bowel syndrome. Gut. 2000 Dec;47(6):804-11. doi: 10.1136/gut.47.6.804. PMID 11076879
- [Background] Pimentel M, Chow EJ, Lin HC. Eradication of small intestinal bacterial overgrowth reduces symptoms of irritable bowel syndrome. Am J Gastroenterol. 2000 Dec;95(12):3503-6. doi: 10.1111/j.1572-0241.2000.03368.x. PMID 11151884
- [Background] Pimentel M, Chow EJ, Lin HC. Normalization of lactulose breath testing correlates with symptom improvement in irritable bowel syndrome. a double-blind, randomized, placebo-controlled study. Am J Gastroenterol. 2003 Feb;98(2):412-9. doi: 10.1111/j.1572-0241.2003.07234.x. PMID 12591062
- [Background] Lupascu A, Gabrielli M, Lauritano EC, Scarpellini E, Santoliquido A, Cammarota G, Flore R, Tondi P, Pola P, Gasbarrini G, Gasbarrini A. Hydrogen glucose breath test to detect small intestinal bacterial overgrowth: a prevalence case-control study in irritable bowel syndrome. Aliment Pharmacol Ther. 2005 Dec;22(11-12):1157-60. doi: 10.1111/j.1365-2036.2005.02690.x. PMID 16305730
- [Background] Cuoco L, Salvagnini M. Small intestine bacterial overgrowth in irritable bowel syndrome: a retrospective study with rifaximin. Minerva Gastroenterol Dietol. 2006 Mar;52(1):89-95. PMID 16554709
- [Background] Majewski M, McCallum RW. Results of small intestinal bacterial overgrowth testing in irritable bowel syndrome patients: clinical profiles and effects of antibiotic trial. Adv Med Sci. 2007;52:139-42. PMID 18217406
- [Background] Shah ED, Basseri RJ, Chong K, Pimentel M. Abnormal breath testing in IBS: a meta-analysis. Dig Dis Sci. 2010 Sep;55(9):2441-9. doi: 10.1007/s10620-010-1276-4. Epub 2010 May 14. PMID 20467896
- [Background] Posserud I, Stotzer PO, Bjornsson ES, Abrahamsson H, Simren M. Small intestinal bacterial overgrowth in patients with irritable bowel syndrome. Gut. 2007 Jun;56(6):802-8. doi: 10.1136/gut.2006.108712. Epub 2006 Dec 5. PMID 17148502
- [Background] Pyleris E, Giamarellos-Bourboulis EJ, Tzivras D, Koussoulas V, Barbatzas C, Pimentel M. The prevalence of overgrowth by aerobic bacteria in the small intestine by small bowel culture: relationship with irritable bowel syndrome. Dig Dis Sci. 2012 May;57(5):1321-9. doi: 10.1007/s10620-012-2033-7. Epub 2012 Jan 20. PMID 22262197
- [Background] Giamarellos-Bourboulis EJ, Pyleris E, Barbatzas C, Pistiki A, Pimentel M. Small intestinal bacterial overgrowth is associated with irritable bowel syndrome and is independent of proton pump inhibitor usage. BMC Gastroenterol. 2016 Jul 11;16(1):67. doi: 10.1186/s12876-016-0484-6. PMID 27402085
- [Background] Pimentel M, Morales W, Pokkunuri V, Brikos C, Kim SM, Kim SE, Triantafyllou K, Weitsman S, Marsh Z, Marsh E, Chua KS, Srinivasan S, Barlow GM, Chang C. Autoimmunity Links Vinculin to the Pathophysiology of Chronic Functional Bowel Changes Following Campylobacter jejuni Infection in a Rat Model. Dig Dis Sci. 2015 May;60(5):1195-205. doi: 10.1007/s10620-014-3435-5. Epub 2014 Nov 26. PMID 25424202
- [Background] Pimentel M, Morales W, Rezaie A, Marsh E, Lembo A, Mirocha J, Leffler DA, Marsh Z, Weitsman S, Chua KS, Barlow GM, Bortey E, Forbes W, Yu A, Chang C. Development and validation of a biomarker for diarrhea-predominant irritable bowel syndrome in human subjects. PLoS One. 2015 May 13;10(5):e0126438. doi: 10.1371/journal.pone.0126438. eCollection 2015. PMID 25970536
- [Background] Shenker BJ, Hoffmaster RH, Zekavat A, Yamaguchi N, Lally ET, Demuth DR. Induction of apoptosis in human T cells by Actinobacillus actinomycetemcomitans cytolethal distending toxin is a consequence of G2 arrest of the cell cycle. J Immunol. 2001 Jul 1;167(1):435-41. doi: 10.4049/jimmunol.167.1.435. PMID 11418680
- [Background] Purdy D, Buswell CM, Hodgson AE, McALPINE K, Henderson I, Leach SA. Characterisation of cytolethal distending toxin (CDT) mutants of Campylobacter jejuni. J Med Microbiol. 2000 May;49(5):473-479. doi: 10.1099/0022-1317-49-5-473. PMID 10798561
- [Background] Pickett CL, Whitehouse CA. The cytolethal distending toxin family. Trends Microbiol. 1999 Jul;7(7):292-7. doi: 10.1016/s0966-842x(99)01537-1. PMID 10390639
- [Background] Eshraghi A, Maldonado-Arocho FJ, Gargi A, Cardwell MM, Prouty MG, Blanke SR, Bradley KA. Cytolethal distending toxin family members are differentially affected by alterations in host glycans and membrane cholesterol. J Biol Chem. 2010 Jun 11;285(24):18199-207. doi: 10.1074/jbc.M110.112912. Epub 2010 Apr 12. PMID 20385557
- [Background] Smith JL, Bayles DO. The contribution of cytolethal distending toxin to bacterial pathogenesis. Crit Rev Microbiol. 2006 Oct-Dec;32(4):227-48. doi: 10.1080/10408410601023557. PMID 17123907
- [Background] Frisk A, Lebens M, Johansson C, Ahmed H, Svensson L, Ahlman K, Lagergard T. The role of different protein components from the Haemophilus ducreyi cytolethal distending toxin in the generation of cell toxicity. Microb Pathog. 2001 Jun;30(6):313-24. doi: 10.1006/mpat.2000.0436. PMID 11399138
- [Background] Torihashi S, Ward SM, Nishikawa S, Nishi K, Kobayashi S, Sanders KM. c-kit-dependent development of interstitial cells and electrical activity in the murine gastrointestinal tract. Cell Tissue Res. 1995 Apr;280(1):97-111. doi: 10.1007/BF00304515. PMID 7538451
- [Background] Rumessen JJ. Ultrastructure of interstitial cells of Cajal at the colonic submuscular border in patients with ulcerative colitis. Gastroenterology. 1996 Dec;111(6):1447-55. doi: 10.1016/s0016-5085(96)70005-7. PMID 8942722
- [Background] Streutker CJ, Huizinga JD, Campbell F, Ho J, Riddell RH. Loss of CD117 (c-kit)- and CD34-positive ICC and associated CD34-positive fibroblasts defines a subpopulation of chronic intestinal pseudo-obstruction. Am J Surg Pathol. 2003 Feb;27(2):228-35. doi: 10.1097/00000478-200302000-00012. PMID 12548170
- [Background] Vanderwinden JM, Liu H, De Laet MH, Vanderhaeghen JJ. Study of the interstitial cells of Cajal in infantile hypertrophic pyloric stenosis. Gastroenterology. 1996 Aug;111(2):279-88. doi: 10.1053/gast.1996.v111.pm8690192.
- [Background] Ordog T, Takayama I, Cheung WK, Ward SM, Sanders KM. Remodeling of networks of interstitial cells of Cajal in a murine model of diabetic gastroparesis. Diabetes. 2000 Oct;49(10):1731-9. doi: 10.2337/diabetes.49.10.1731. PMID 11016458
- [Background] Bassotti G, Villanacci V, Maurer CA, Fisogni S, Di Fabio F, Cadei M, Morelli A, Panagiotis T, Cathomas G, Salerni B. The role of glial cells and apoptosis of enteric neurones in the neuropathology of intractable slow transit constipation. Gut. 2006 Jan;55(1):41-6. doi: 10.1136/gut.2005.073197. Epub 2005 Jul 24. PMID 16041063
- [Background] Pimentel M, Chatterjee S, Chow EJ, Park S, Kong Y. Neomycin improves constipation-predominant irritable bowel syndrome in a fashion that is dependent on the presence of methane gas: subanalysis of a double-blind randomized controlled study. Dig Dis Sci. 2006 Aug;51(8):1297-301. doi: 10.1007/s10620-006-9104-6. Epub 2006 Jul 11. PMID 16832617
- [Background] Sharara AI, Aoun E, Abdul-Baki H, Mounzer R, Sidani S, Elhajj I. A randomized double-blind placebo-controlled trial of rifaximin in patients with abdominal bloating and flatulence. Am J Gastroenterol. 2006 Feb;101(2):326-33. doi: 10.1111/j.1572-0241.2006.00458.x. PMID 16454838
- [Background] Pimentel M, Park S, Mirocha J, Kane SV, Kong Y. The effect of a nonabsorbed oral antibiotic (rifaximin) on the symptoms of the irritable bowel syndrome: a randomized trial. Ann Intern Med. 2006 Oct 17;145(8):557-63. doi: 10.7326/0003-4819-145-8-200610170-00004. PMID 17043337
- [Background] Pimentel M, Lembo A, Chey WD, Zakko S, Ringel Y, Yu J, Mareya SM, Shaw AL, Bortey E, Forbes WP; TARGET Study Group. Rifaximin therapy for patients with irritable bowel syndrome without constipation. N Engl J Med. 2011 Jan 6;364(1):22-32. doi: 10.1056/NEJMoa1004409. PMID 21208106
- [Background] Debbia EA, Maioli E, Roveta S, Marchese A. Effects of rifaximin on bacterial virulence mechanisms at supra- and sub-inhibitory concentrations. J Chemother. 2008 Apr;20(2):186-94. doi: 10.1179/joc.2008.20.2.186. PMID 18467244
- [Background] Jiang ZD, DuPont HL. Rifaximin: in vitro and in vivo antibacterial activity--a review. Chemotherapy. 2005;51 Suppl 1:67-72. doi: 10.1159/000081991. PMID 15855749
- [Background] Gerard L, Garey KW, DuPont HL. Rifaximin: a nonabsorbable rifamycin antibiotic for use in nonsystemic gastrointestinal infections. Expert Rev Anti Infect Ther. 2005 Apr;3(2):201-11. doi: 10.1586/14787210.3.2.201. PMID 15918778
- [Background] Fodor AA, Pimentel M, Chey WD, Lembo A, Golden PL, Israel RJ, Carroll IM. Rifaximin is associated with modest, transient decreases in multiple taxa in the gut microbiota of patients with diarrhoea-predominant irritable bowel syndrome. Gut Microbes. 2019;10(1):22-33. doi: 10.1080/19490976.2018.1460013. Epub 2018 Jul 18. PMID 29708822
- [Background] Pimentel M, Lembo A. Microbiome and Its Role in Irritable Bowel Syndrome. Dig Dis Sci. 2020 Mar;65(3):829-839. doi: 10.1007/s10620-020-06109-5. PMID 32026278
- [Background] Mearin F, Lacy BE, Chang L, Chey WD, Lembo AJ, Simren M, Spiller R. Bowel Disorders. Gastroenterology. 2016 Feb 18:S0016-5085(16)00222-5. doi: 10.1053/j.gastro.2016.02.031. Online ahead of print. PMID 27144627
- [Derived] Villanueva-Millan MJ, Leite G, Wang J, Morales W, Parodi G, Pimentel ML, Barlow GM, Mathur R, Rezaie A, Sanchez M, Ayyad S, Cohrs D, Chang C, Rashid M, Hosseini A, Fiorentino A, Weitsman S, Chuang B, Chang B, Pichetshote N, Pimentel M. Methanogens and Hydrogen Sulfide Producing Bacteria Guide Distinct Gut Microbe Profiles and Irritable Bowel Syndrome Subtypes. Am J Gastroenterol. 2022 Dec 1;117(12):2055-2066. doi: 10.14309/ajg.0000000000001997. Epub 2022 Sep 6. PMID 36114762
- [Derived] Pimentel M, Mathur R, Wang J, Chang C, Hosseini A, Fiorentino A, Rashid M, Pichetshote N, Basseri B, Treyzon L, Chang B, Leite G, Morales W, Weitsman S, Kraus A, Rezaie A. A Smartphone Application Using Artificial Intelligence Is Superior To Subject Self-Reporting When Assessing Stool Form. Am J Gastroenterol. 2022 Jul 1;117(7):1118-1124. doi: 10.14309/ajg.0000000000001723. Epub 2022 Mar 14. PMID 35288511

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Dose for IBS-D | Traveler's Diarrhea Dose + Placebo | Traveler's Diarrhea Dose + NAC
Started | 15 | 15 | 15
Completed | 15 | 15 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Dose for IBS-D | Traveler's Diarrhea Dose + Placebo | Traveler's Diarrhea Dose + NAC | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 15 | 45
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (17) | 44 (14) | 47 (13) | 45.89 (15.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 7 | 29
  Male | 5 | 3 | 8 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 14 | 12 | 13 | 39
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 15 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change in Stool Form
Description: Change in stool form from baseline, as determined from stool diary data comparing Rifaximin alone vs rifaximin and NAC
  The Bristol Stool Chart, the minimum value is 1 (means constipation) and maximum value is 7 (means diarrhea).
  The change between two time points is reported baseline and 4 weeks after cessation of treatment (at 6 weeks)
Time Frame: value at 6 weeks minus value at baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Rifaximin 550 mg: Rifaximin 550 mg Standard dose for IBS-D
  Rifaximin: Rifaximin is indicated for the treatment of irritable bowel syndrome with diarrhea (IBS-D) in adults.
- Rifaximin 200 mg + Placebo: Rifaximin 200 mg + placebo Traveler's diarrhea dose + placebo
  Rifaximin: Rifaximin is indicated for the treatment of irritable bowel syndrome with diarrhea (IBS-D) in adults.
  Placebo: An inactive substance or treatment that looks the same as, and is given in the same way as, an active drug or intervention/treatment being studied.
- Rifaximin 200 mg Plus N-acetylcysteine (NAC) 600 mg Days: Rifaximin 200 mg plus N-acetylcysteine (NAC) 600 mg days Traveler's diarrhea dose + NAC
  Rifaximin: Rifaximin is indicated for the treatment of irritable bowel syndrome with diarrhea (IBS-D) in adults.
  N-acetylcysteine: N-acetylcysteine (NAC) is a clinically approved mucolytic agent.
Arm/Group | Rifaximin 550 mg | Rifaximin 200 mg + Placebo | Rifaximin 200 mg Plus N-acetylcysteine (NAC) 600 mg Days
Number analyzed (Participants) | 15 | 15 | 15
score on a scale | -0.26 (0.69) | -0.45 (0.86) | -0.49 (0.72)

2. Primary Outcome: Change in Abdominal Pain
Description: Change in severity of abdominal pain from baseline, as determined from weekly average visual analog scale (VAS) scores, relative to Rifaximin alone. VAS scores allows subject to choose 0 for "no pain" to 100 "pain as bad as it could possibly be".
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 "no pain" and 100 "pain as bad as it could possibly be"
  The change between two time points is reported baseline and 4 weeks after cessation of treatment (at 6 weeks)
Time Frame: value at 6 weeks minus value at baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Rifaximin 550 mg: Standard dose for IBS-D
  Rifaximin: Rifaximin is indicated for the treatment of irritable bowel syndrome with diarrhea (IBS-D) in adults.
- Rifaximin 200 mg + Placebo: Traveler's diarrhea dose + placebo
  Rifaximin: Rifaximin is indicated for the treatment of irritable bowel syndrome with diarrhea (IBS-D) in adults.
  Placebo: An inactive substance or treatment that looks the same as, and is given in the same way as, an active drug or intervention/treatment being studied.
- Rifaximin 200 mg Plus N-acetylcysteine (NAC) 600 mg Days: Traveler's diarrhea dose + NAC
  Rifaximin: Rifaximin is indicated for the treatment of irritable bowel syndrome with diarrhea (IBS-D) in adults.
  N-acetylcysteine: N-acetylcysteine (NAC) is a clinically approved mucolytic agent.
Arm/Group | Rifaximin 550 mg | Rifaximin 200 mg + Placebo | Rifaximin 200 mg Plus N-acetylcysteine (NAC) 600 mg Days
Number analyzed (Participants) | 15 | 15 | 15
units on a scale | -5.43 (13.91) | -8.90 (21.42) | -5.59 (15.99)

3. Primary Outcome: Change in Stool Frequency
Description: Change in stool frequency from baseline, as determined from diary data comparing Rifaximin alone vs Rifaximin and NAC
  determined from daily stool diary data
  The change in bowel movements/day between two time points is reported baseline and 4 weeks after cessation of treatment (at 6 weeks)
Time Frame: value at 6 weeks minus value at baseline
Measure: Mean (Standard Deviation); unit: number of bowel movements
Groups:
- Rifaximin 550 mg: Rifaximin 550 mg (Standard dose for IBS-D)
  Rifaximin: Rifaximin is indicated for the treatment of irritable bowel syndrome with diarrhea (IBS-D) in adults.
- Rifaximin 200 mg + Placebo: Rifaximin 200 mg + placebo (Traveler's diarrhea dose + placebo)
  Rifaximin: Rifaximin is indicated for the treatment of irritable bowel syndrome with diarrhea (IBS-D) in adults.
  Placebo: An inactive substance or treatment that looks the same as, and is given in the same way as, an active drug or intervention/treatment being studied.
- Rifaximin 200 mg Plus N-acetylcysteine (NAC) 600 mg Days: Traveler's diarrhea dose + NAC (Rifaximin 200 mg plus N-acetylcysteine (NAC) 600 mg days)
  Rifaximin: Rifaximin is indicated for the treatment of irritable bowel syndrome with diarrhea (IBS-D) in adults.
  N-acetylcysteine: N-acetylcysteine (NAC) is a clinically approved mucolytic agent.
Arm/Group | Rifaximin 550 mg | Rifaximin 200 mg + Placebo | Rifaximin 200 mg Plus N-acetylcysteine (NAC) 600 mg Days
Number analyzed (Participants) | 15 | 15 | 15
number of bowel movements | -0.04 (0.64) | -0.50 (1.50) | -0.24 (0.80)

ADVERSE EVENTS:
Time Frame: 6 weeks
Groups:
- Rifaximin 200 mg Plus N-acetylcysteine (NAC) 600 mg Days: Rifaximin 200 mg plus N-acetylcysteine (NAC) 600 mg days (Traveler's diarrhea dose + NAC)
  Rifaximin: Rifaximin is indicated for the treatment of irritable bowel syndrome with diarrhea (IBS-D) in adults.
  N-acetylcysteine: N-acetylcysteine (NAC) is a clinically approved mucolytic agent.
Arm/Group | Rifaximin 550 mg | Rifaximin 200 mg + Placebo | Rifaximin 200 mg Plus N-acetylcysteine (NAC) 600 mg Days
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 2/15 | 2/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rifaximin 550 mg (N=15) | Rifaximin 200 mg + Placebo (N=15) | Rifaximin 200 mg Plus N-acetylcysteine (NAC) 600 mg Days (N=15)
Bloating & Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea and vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Headache and nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Burning in esophagus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-10): https://cdn.clinicaltrials.gov/large-docs/15/NCT04557215/Prot_SAP_000.pdf